CLINICAL TRIAL: NCT05992636
Title: The Effects of Hemodynamic Changes on Cerebral Oxygenation Caused by Pneumoperitoneum With Different Insufflation Flows in Laparoscopic Cholecystectomy
Brief Title: Different Insufflation Flows and Effects on Cerebral Oxygenation in Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, SEDAT SAYLAN, Associate Prof., Karadeniz Technical University
Other Study IDs: Karadeniz Teknik Üniversitesi
Record Dates: First submitted 2021-11-12; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Pneumoperitoneum
Keywords: laparoscopic cholecystectomy; Near Infrared Spectroscopy (NIRS)
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- low insufflation flow (10 lt/min): Patiens who perform pneumoperitoneum with low insufflation flow (10 lt/min)
  Interventions: Procedure: pneumoperitoneum insufflation (flow) rate
- high insufflation flow (40 lt/min): Patiens who perform pneumoperitoneum with high insufflation flow (40 lt/min)
  Interventions: Procedure: pneumoperitoneum insufflation (flow) rate

INTERVENTIONS:
Procedure: pneumoperitoneum insufflation (flow) rate — Patiens who initiate with low insufflation flow (10 lt/min)
  Patiens who initiate with high insufflation flow (40 lt/min)

SUMMARY:
Previous studies conducted on the hemodynamic effects of pneumoperitoneum pressures created by different insufflation flows are very limited in the literature. In a current literature review, there was no study found comparing the effects of hemodynamic changes created by low and high insufflation flows and pneumoperitoneum pressure on cerebral oxygenation. The purpose of the study was to contribute to the literature by investigating the effects of pneumoperitoneum pressures created by different flows on brain oxygenation.

DETAILED DESCRIPTION:
After the approval of the Ethics Committee, a total of 69 (sixty-nine) patients who would undergo elective laparoscopic cholecystectomy were planned as ASA I-III, 18-65 years old, 34 (thirty-four) patients low insufflation flow (10 lt/min) and 35 (thirty-five) patients and high insufflation flow (40 lt/min) with pneumoperitoneum pressure.

The study will be conducted as a single-center observational study in Trabzon KTU Faculty of Medicine General Surgery Operating Room. Anesthesia always be performed by the same anesthesia team, and no intervention will be made regarding the choice of the method. The data obtained will be recorded by the anesthetists other than the team who constitute the study group, and the data obtained at the end of the surgery will be interpreted by the study team. The decision for laparoscopic cholecystectomy of the patients who will be included in the study will be made by the General Surgery doctor, and the patients who are scheduled to be operated on electively will be included in the study.

The patients will be taken to the operating room after their written consents are obtained and preoperative evaluations are made, and routine premedication will be applied to the patients who arrive at the operating room. The patients who will be included in the study will be monitored routinely in the general surgery room (i.e. electrocardiography (ECG), non-invasive blood pressure measurement, peripheral oxygen saturation, Bispectral Index (BIS), and additionally NIRS monitoring. No interference will be made regarding the groups in which patients who will undergo general anesthesia will be in the pneumoperitoneum group formed with low insufflation flow or high insufflation flow, only non-invasive cerebral oxygenation measurements will be made with NIRS monitor (INVOS™ 5100C Cerebral/Somatic Oximeter, SOMANETICS, COVIDIEN, Mansfield/ USA)

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy were planned,
* ASA I-III,
* 18-65 years old

Exclusion Criteria:

* Cerebrovascular diseases and/or intracranial pathologies and/or related neurological events,
* Uncontrolled diabetes
* Uncontrolled hypertension
* Coagulopathy,
* Cirrhosis and/or peritonitis,
* Asthma and/or respiratory diseases e.g. COPD,
* Morbid obesity,
* Patients with severe organ failure,
* Emergency cases,
* Cases converted to laparotomic cholecystectomy.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After the approval of the Ethics Committee, a total of 69 (sixty) patients who would undergo elective laparoscopic cholecystectomy were planned as ASA I-III, 18-65 years old, 34 (thirty-four) patients with low insufflation flow (10 lt/min), and 35 (thirty-five) patients in high insufflation flow (40 lt/min) with pneumoperitoneum pressure.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
the relationship between insufflation flow rate and cerebral desaturation (rSO2) | 8 months
  With this study, the results of hemodynamic effects on cerebral oxygenation caused by two different insufflation flows (10 lt/min and 40 lt/min) was evaluated by used to create iatrogenic pneumoperitoneum in laparoscopic cholecystectomy surgery with a non-invasive technique, Near Infrared Spectroscopy (NIRS).
  The primary outcome is the investigate to relationship between insufflation flow rate and cerebral desaturation ( which defined by 20% or more decrease in cerebral oxygen saturation compared to baseline value of the patient )

SECONDARY OUTCOMES:
the relationship between insufflation flow rate and end-tidal carbon dioxide value variation (mmHg) | 8 months
  Relationship between insufflation flow rate and end-tidal carbon dioxide value variation of the patients according to basal and before-pnömoperitoneum end-tidal carbon dioxide levels (mmHg) was determined with capnographic measurements.
the relationship between insufflation flow rate and heart rate value variation (beats per minute) | 8 months
  Relationship between insufflation flow rate and heart rate value variation of the patients according to basal and before-pnömoperitoneum heart rate levels was determined with pulse monitoring.
the relationship between insufflation flow rate systolic, diastolic and mean arterial pressure values variation (mmHg) | 8 months
  Relationship between insufflation flow rate and systolic, diastolic and mean arterial pressure (mmHg) values variation of the patients according to basal and before-pnömoperitoneum systolic, diastolic and mean arterial pressure levels were determined with non-invasive blood pressure measurements.

CONTACTS AND LOCATIONS:
Overall Officials: KIVANÇ ÖNCÜ, M.D., Study Chair — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)